CLINICAL TRIAL: NCT06521632
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Cognitive Function Under Exposure to Hypoxia
Brief Title: Acupoint Stimulation Improves Cognition Under Hypoxia
Acronym: TREACLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhihong LU (Other)
Responsible Party: Sponsor-Investigator, Zhihong LU, Associate professor, Air Force Military Medical University, China
Organization: Air Force Military Medical University, China (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: XJH-A-20240319
Record Dates: First submitted 2024-07-04; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Cognition
Keywords: transcutaneous electrical acupoint stimulation; cognition; hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The stimulator is put in an opaque box
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transcutaneous electrical acupoint stimulation (Experimental): Electrodes are placed at acupoints and connected to the stimulators. Electrical stimulation is given for 2 hours
  Interventions: Other: transcutaneous electrical acupoint stimulation
- Control (No Intervention): Electrodes are placed at acupoints but no electrical stimulation is given

INTERVENTIONS:
Other: transcutaneous electrical acupoint stimulation — Electrodes are placed at acupoints and connected to the stimulator. Electrical stimulation is given for 2 hours.
  Arms: transcutaneous electrical acupoint stimulation

SUMMARY:
Cognitive impairment is common in people who suffer from hypoxia. Acupuncture and related techniques can be used to improve hypoxia and treat cognitive impairment. In this trial the effect of transcutaneous electrical acupoint stimulation on cognitive impairment in people under hypoxia will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male, age from 18 to 50 years

Exclusion Criteria:

* cardiopulmonary dysfunction;
* History of severe respiratory, circulatory, digestive, blood, ear-nose-throat system diseases;
* A history of fever or respiratory infection within the last two weeks;
* Drinking alcohol or poor sleep within the last 24 hours

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-07 (Estimated)

PRIMARY OUTCOMES:
cognitive function measured by eye-tracking at 1 hour after hypoxia | 1 hour after hypoxia
cognitive function measured by eye-tracking at 2 hours after hypoxia | 2 hours after hypoxia

SECONDARY OUTCOMES:
mean arterial blood pressure | starting from 10 minutes before hypoxia to 2 hours after hypoxia, every 5 minutes for 2 hours and 10 minutes
heart rate | starting from 10 minutes before hypoxia to 2 hours after hypoxia, every 5 minutes for 2 hours and 10 minutes
saturation of pulse oximetry | starting from 10 minutes before hypoxia to 2 hours after hypoxia, every 5 minutes for 2 hours and 10 minutes
Cerebral oxygen saturation | starting from 10 minutes before hypoxia to 2 hours after hypoxia, every 5 minutes for 2 hours and 10 minutes
total sleep time on the first day after hypoxia | the first day after hypoxia, in a total of 24 hours
sleep efficiency(%) on the first day after hypoxia | the first day after hypoxia, in a total of 24 hours
  sleep efficiency=total sleep time/total recording time
number of awake on the first day after hypoxia | the first day after hypoxia, in a total of 24 hours
time of awake on the first day after hypoxia | the first day after hypoxia, in a total of 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No